CLINICAL TRIAL: NCT05048173
Title: Sentinel Lymph Node Biopsy Versus Pelvic Lymphadenectomy in Early Stage Endometrial Cancer
Brief Title: Sentinel Lymph Node Biopsy Versus Lymphadenectomy in Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 110187-E
Record Dates: First submitted 2020-12-18; First posted 2021-09-17 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Early Stage Endometrial Cancer; Sentinel Lymph Nodes; Lymphadenectomy
MeSH Terms: interventions — Biopsy; Lymph Node Excision

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sentinel lymph node group: woman who had sentinel lymph node mapping and biopsy
  Interventions: Procedure: Sentinel lymph node mapping and biopsy
- Lymphadenectomy group: woman who underwent traditional pelvic lymphadenectomy without sentinel lymph node mapping
  Interventions: Procedure: Lymphadenectomy

INTERVENTIONS:
Procedure: Sentinel lymph node mapping and biopsy — Sentinel lymph node mapping with indocyanine green dye followed by biopsy if positive
  Groups: Sentinel lymph node group
Procedure: Lymphadenectomy — Conventional lymphadenectomy
  Groups: Lymphadenectomy group

SUMMARY:
To compare sentinel lymph nodes biopsy versus comprehensive lymphadenectomy in patients with early stage endometrial cancer.

DETAILED DESCRIPTION:
This retrospective study aims to compare sentinel lymph nodes biopsy versus comprehensive lymphadenectomy in patients with early stage endometrial cancer by reviewing the medical records.

ELIGIBILITY:
Inclusion Criteria:

* ≧ 20 years
* early stage endometrial cancer (FIGO stage I)

Exclusion Criteria:

* Did not receive a complete course of treatment in this hospital, interrupted the treatment halfway (except if the disease continued to deteriorate or caused death during treatment), and did not follow up in this hospital after the course of treatment.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — early stage endometrial cancer
Study Population: Women aged 20 and above, diagnosed with early stage endometrial cancer (FIGO stage I), who had received staging surgery between 01 July 2017 and 19 August 2021 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
progression free survival | 4 years
  The length of time from the day of operation till recurrence or last follow up
overall survival | 4 years
  The length of time from the day of operation till death (of any cause) or last follow up

SECONDARY OUTCOMES:
surgical complications related to lymph node biopsy or lymphadenectomy | from the day of operation till post-operative 6 months
  asymptomatic lymphocele, lymphedema, infected lymphocele

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan